CLINICAL TRIAL: NCT02005068
Title: Ceftaroline in the Treatment of Bone and Joint Infections
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Failed to enroll any patients despite study modifications
Sponsor: Orlando Health, Inc. (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Mark Wallace MD, Infectious Disease Faculty Practice, Orlando Health, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TEF-IT-17
Record Dates: First submitted 2013-11-21; First posted 2013-12-09 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Osteomyelitis; Joint Infections
Keywords: Osteoarticular infections; Osteomyelitis; Joint infections; MRSA (Methicillin- Resistant Staphylococcus Aureus); MSSA (Methicillin- Susceptible Staphylococcus Aureus)
MeSH Terms: conditions — Osteomyelitis | interventions — Ceftaroline; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Acute Osteomyelitis - Non MRSA (Experimental): For treatment of Acute osteomyelitis (< 6 months duration) Non MRSA isolate- Ceftaroline 600 MG (milligram) IV (intra-venous) every 8 hours for 6 weeks.
  Interventions: Drug: Ceftaroline
- Acute osteomyelitis MRSA isolate (Experimental): For treatment of Acute osteomyelitis (< 6 months duration) MRSA isolate- Ceftaroline 600 MG IV every 8 hours for 8 weeks.
  Interventions: Drug: Ceftaroline
- Prosthetic joint infection (Experimental): For treatment of prosthetic joint infection Ceftaroline 600 mg IV every 8 hours for 6 weeks.
  Interventions: Drug: Ceftaroline

INTERVENTIONS:
Drug: Ceftaroline — The duration of treatment will vary based on type of infection (acute osteomyelitis or joint infection) and if MRSA positive or negative.
  Other Names: Teflaro; Ceftaroline fosamil; PPI-0903; TAK-599,; ceftaroline acetate; ceftaroline prodrug; ceftaroline fosamil for injection; Ceftaroline: PPI-0903M; T 91825; Chemical Name (6R,7R)-7-{(2Z)-2-(ethoxyimino)-2-[5-; (phosphonoamino)-1,2,4-thiadiazol-3-; yl]acetamino}-3-[(4-(1-methylpyridin-1-ium-4-yl)-; 1,3-thiazol-2-yl]sulfanyl}-8-oxo-5-thia-1-; azabicyclo[4.2.0]oct-2-ene-2-carboxylate

SUMMARY:
This is a study to evaluate the efficacy of Ceftaroline in the treatment of bone and joint infections.

DETAILED DESCRIPTION:
Study evaluates the efficacy of Ceftaroline 600mg IV every 8 hours for the treatment of acute osteomyelitis and/or infected joints.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years of age with the following osteoarticular infections:

  1. Infected prosthetic knee or hip (first or second episode) with 2 stage procedure planned.

     Criteria for infected joint:
     1. Sinus tract which communicates with the joint
     2. Preoperative diagnosis by diagnostic, culture positive arthrocentesis
     3. Intraoperative diagnosis-evidence of purulence/inflammation is seen by the surgeon and/or the pathologist, and at least 2 intraoperative samples grow the same organism (only 1 needed if S. aureus) OR
  2. Acute osteomyelitis of an extremity Criteria for acute osteomyelitis (all 4 needed)

     1. Onset less than 4 weeks prior to evaluation
     2. Radiographic (plain, MRI, TC) evidence of osteomyelitis
     3. Positive culture from bone or blood culture with organism known to cause osteomyelitis
     4. Orthopedic consultant must concur with diagnosis. PLUS: Positive bone/joint or blood culture for an organism known to cause osteomyelitis which is Ceftaroline susceptible

Exclusion criteria:

1. Immunocompromised hosts:

   1. AIDS/HIV patients
   2. Cancer requiring ongoing chemotherapy or radiation therapy steroid on an ongoing basis.
   3. Any condition requiring > 20 mg prednisone or equivalent
   4. TNF (tumor necrosing factor) inhibitor use (ongoing)
   5. Organ transplant list
2. Diabetic foot infections
3. Osteomyelitis in association with decubitus ulcers
4. Vertebral osteomyelitis/spinal epidural abscess
5. Septic bursitis
6. Gonococcal arthritis
7. Ceftaroline nonsusceptible organisms isolated from bone, joint or blood.
8. Infected external fixation devices
9. Calculated creatinine clearance < 50 mL/min at baseline
10. History of severe penicillin/B lactam allergy (ID to evaluate)
11. Intravenous drug use - lifetime exclusion
12. Patients with a nail puncture wound to foot
13. Patients at high risk for MDR (multidrug resistant) Gram negative organisms

Please note the use of antibiotic containing cement is not exclusion, as it represents standard of care in some of the infections to be studied

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Sustained clinical remission from the treated osteoarticular infection | 1 year after study drug completion
  Sustained clinical remission is defined by the absence of either clinical or microbiological evidence of failure at 1 year after study drug completion, in patients who complete the protocol's antibiotic regimen(s) and did not require subsequent antibiotics for their osteoarticular infection beyond the protocol prescribed regimen.

SECONDARY OUTCOMES:
Initial clinical success from the treated osteoarticular infection | 30 days after conclusion of study antibiotic
  Initial clinical success will be measured by the agreement of the Infectious disease consultant and Orthopedic surgeon that the patient has had a positive response to therapy. Success will be measured by decrease of CRP (C reactive protein) by 50% from baseline if initially elevated, no evidence of drainage, sinus tract formation or infection related bone instability. Follow up cultures, if available are negative for originally isolated organism. In patients with prothetic joints no new warmth, tenderness or inflammation.

OTHER OUTCOMES:
Number of participants with defined symptoms, signs and lab values as markers of safety and tolerance. | Day one through one year after completion of study drug.
  Symptoms will be assessed daily by study team while patient is hospitalized and reviewed weekly by investigator while the patient is receiving study drug. Specific symptoms will include fever, chills, rash, nausea. diarrhea, abdominal pain, pain at the surgical/infection site, vertigo, shortness of breath, hives or other rash. A baseline physical will be performed on enrollment and repeated each week at follow up visits. Labs will checked at baseline, then daily through hospitalization and then weekly. If patient develops persistent diarrhea a stool test for C. Diff PCR (polymerase chain reaction) will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Mark R. Wallace, MD, Principal Investigator — Orlando Health
Locations (1):
- Orlando Regional Medical Center, Orlando, Florida, United States